CLINICAL TRIAL: NCT04715672
Title: The Establishment of Evaluation Model About Returning to Sports Post-operation of Anterior Cruciate Ligament Reconstruction by Resting State Functional Magnetic Resonance and Three-dimensional Gait Analysis
Brief Title: The Establishment of Advanced Brain Function Evaluation Model for Anterior Cruciate Ligament Reconstruction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-144
Record Dates: First submitted 2021-01-13; First posted 2021-01-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Anterior Cruciate Ligament Reconstruction;Resting State Functional Magnetic Resonance;Three-dimensional Gait Analysis;Return to Sports

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- copper
- no-copper
- normal

SUMMARY:
It is difficult to establish the standard of return to sports post anterior cruciate ligament (ACL) reconstruction. The amplitude of low frequency fluctuation (ALFF) and functional connectivity (FC) of resting state functional magnetic resonance imaging (fMRI) can explore the differences in neural function of different populations, but have not been applied in the study of ACL postoperative return to sports.This project intends to use ALFF algorithm to calculate the changes of BLOD signals of coppers and non- coppers after ACL surgery in the subfrequency band and the functional network in the subfrequency band, explore the relationship between the default network (DMN) and the sensorimotor network (SMN), and use three-dimensional gait analysis to carry out accurate functional test..This project will explore the central strategy of ACL postoperative functional recovery from a new perspective, to provide a more reasonable high-level evaluation index for the timing of return to sports, and to reduce the incidence of postoperative re-tearing.

ELIGIBILITY:
Inclusion Criteria:

Patients who completed the same operation and completed phased home rehabilitation instruction and who underwent ACL reconstruction more than 2 years after the operation were recruited as the test subjects

Exclusion Criteria:

heart and nervous system diseases, Other sports injuries such as medial collateral ligament injury, meniscus repair, grade III-IV cartilage injury, ankle instability, metal implants in the body and medication were excluded

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: patients post anteriorcruciate ligament (ACL) reconstruction
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
ALFF | 2 years post-operation
  ALFF algorithm to calculate BLOD signals in the subfrequency band of resting state functional magnetic resonance imaging (fMRI)
FC | 2 years post-operation
  functional connection between brain region of interest in the subfrequency band of resting state magnetic resonance imaging (fMRI)

SECONDARY OUTCOMES:
Lysholm | 2 years post-operation
  Lysholm scale, which is used to measure the functional status of a patient's knee joint has a minimum value of 0 and a maximum value of 100, with the higher the score, the better the function
Tegner | 2 years post-operation
  Tegner scale，which is used to measure the functional status of patients has a minimum value of 0 and a maximum value of 10, with the higher the score, the better of the function.
COP（center of pressure ） | 2 years post-operation
  symmetry of center of pressure transfer path by using Plantar pressure testing system when patients are walking and running. limb symmetry index =injury limb score/good limb score *100
CR | 2 years post-operation
  Hamstring Co-contraction ratio(CR) in the Single foot support phase by using the Surface electromyography when patients are walking and running.
single leg jump test | 2 years post-operation
  Patient stands onhis or her leg , toe on starting line, try to jump forward and land on ipsilateral limb, measure the distance between starting line and patient's feet. limb symmetry index =injury limb score/good limb score *100
6M timing single leg jump test | 2 years post-operation
  The patient stood on his or her leg, with the toes on the starting line. After the tester gave the command of "each in position, prepare, run", the chronograph was accurate to 0.01 seconds to start the time. The patient's healthy limbs jump as soon as possible and stop the timing when reaching the 6m terminal.limb symmetry index =injury limb score/good limb score *100

CONTACTS AND LOCATIONS:
Locations (1):
- Hongyun song, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR